CLINICAL TRIAL: NCT05387434
Title: The National Diabetes Prevention Program in Rural Communities
Acronym: Rural NDPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Kansas State University (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00146055; 5P20GM144269 (NIH)
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: PreDiabetes; Weight Loss; Lifestyle Risk Reduction
MeSH Terms: conditions — Prediabetic State; Weight Loss; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: The proposed 2-arm trial will compare the feasibility and effectiveness of Facebook or remote-delivery of the DPP in rural adults with prediabetes both delivered through the KSRE. The CES is a non-formal educational program, implemented in the U.S. through each state's designated land grant university, to help people use research-based knowledge to improve their lives. The KSRE maintains local units which are comprised of single counties or multi-county districts. Two KSRE local units serving rural counties will be identified by our partners at KSRE and randomized to the Facebook or remote delivery arms. Members of the KUMC research team will recruit and consent participants and will train KSRE personnel to deliver the 30 core-sessions of the DPP protocol over 12 mos. Outcomes will be assessed by the research team at the local CES offices at baseline, 3 mos. 6 mos. and 12 mos.
Who Masked: Participant
Masking Description: Two rural KSRE local units will be randomized in a 1:1 ratio to either DPP-FB or DPP-R.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPP-R (Experimental): Weekly 60 min. group meetings, lead by trained KSRE staff, (12-15 participants) will be held by Zoom over 6 months followed by monthly 60 min. group meetings for the later 6 months. Approximately 5 min prior to the meeting time (typically early evening) participants will receive call in information to join the group meeting by video conferencing or phone.
  Interventions: Behavioral: Diabetes Prevention Program-Remote (DPP-R)
- DPP-FB (Experimental): Participants will be asked to join a secret, research team moderated, Facebook® group, which is only accessible by group members. The health educator will post the module, de-identified participant self-monitoring data, and comment on individuals posts weekly. Brief discussion prompts are designed to reinforce the primary objectives of each module and to facilitate inter-participant discussion around these topics. Responses will be monitored and tracked. This is analogous to attendance in the Zoom® group.
  Interventions: Behavioral: Diabetes Prevention Program-Facebook (DPP-FB)

INTERVENTIONS:
Behavioral: Diabetes Prevention Program-Remote (DPP-R) — The DPP is an evidenced based lifestyle intervention that includes topics on nutrition and physical activity delivered over Zoom.
  Arms: DPP-R
Behavioral: Diabetes Prevention Program-Facebook (DPP-FB) — The DPP is an evidenced based lifestyle intervention that includes topics on nutrition and physical activity delivered over Facebook.
  Arms: DPP-FB

SUMMARY:
The purpose of this pilot trial is to compare feasibility and effectiveness of remote delivery (social media or video conferencing) of the National Diabetes Prevention Program (N-DPP) to adults in rural communities. The research team will train a Kansas State Research and Extension staff to deliver the video conferencing arm while a research team member will lead the social media arm.

DETAILED DESCRIPTION:
This pilot trial will compare the feasibility and effectiveness of DPP delivered through Facebook (DPP-FB) or group format delivered remotely by Zoom (DPP-R) in adults in rural communities. Both interventions will recruit through the Corporative Extension Service (CES), which serves as the community outreach arm of all land grant universities through over 2,900 offices across the U.S. The Kansas State Research and Extension (KSRE) (Kansas version of CES), is well positioned, but underutilized for the delivery of DPP in rural areas. Delivery of DPP by a well-recognized entity, such as the KSRE, may improve the probability of dissemination and long-term program sustainability. Two CES offices serving rural counties in Kansas will be randomized (1:1) to the DPP-FB or DPP-R arms. Our research team will train one professional staff from KSRE (with backgrounds in nutrition programming and family consumer science) to deliver the DPP-R intervention. A research team member will deliver the DPP-FB intervention. This project will address the following aims:

Primary aim: Compare weight and MVPA between DPP-FB and DPP-R across 6 mos. The investigators expect greater weight loss and MVPA in the DPP-R arm compared with the DPP-FB arm.

Secondary aim: Compare the feasibility of DPP-FB and DPP-R across 6 mos. based on participant retention and program attendance. The investigators expect greater participant retention and program attendance in the DPP-R arm compared with the DPP-FB arm.

ELIGIBILITY:
Inclusion Criteria:

1. Prediabetes as defined as A1C = 5.7-6.4%, fasting glucose = 100-125 mg/dl, (confirmed from physician/medical record in the previous year), history of gestation diabetes mellitus OR a positive result based on the CDC- DPP screener
2. Age ≥18 yrs.
3. Willing to commit to participate on a weekly basis for the 6 month intervention
4. Living in the county of a rural KSRE local unit. Rural counties will be defined using the American Community Survey definition which categorizes a county as rural if the population is < 65,000
5. Internet access and capability to use Zoom
6. Clearance from primary care physician

Exclusion Criteria:

1. Diagnosis of Type 2 diabetes
2. Unable to participate in physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Gorczyca, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wagner G, Koon LM, Smith P, Suire KB, Hastert M, Donnelly JE, Olfert MD, Estabrooks P, Gorczyca AM. Assessing the Fit of a Digitally Delivered National Diabetes Prevention Program Among Rural Living Adults: Qualitative Study. JMIR Form Res. 2025 Jul 2;9:e70406. doi: 10.2196/70406. PMID 40601375

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DPP-R | DPP-FB
Started | 16 | 15
Completed | 14 | 13
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DPP-R | DPP-FB | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (11.1) | 53.8 (14.7) | 55.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight From 0-6 Months
Description: Anthropometric measurements: Body weight will be assessed to the nearest 0.1 kg with a calibrated scale (Belfour Inc., Model #PS6600, Saukville, WI). All participants will be weighed between the hours of 6 and 11 am following a 12 hr. fast in a standard hospital gown.
Time Frame: Baseline - 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | DPP-R | DPP-FB
Number analyzed (Participants) | 14 | 13
kilograms | -6.0 (8.0) | -1.7 (3.3)

2. Secondary Outcome: Participant Retention
Description: Retention will be defined as attendance at 6 mo. outcome testing.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DPP-R | DPP-FB
Number analyzed (Participants) | 16 | 15
Participants | 14 | 13

3. Secondary Outcome: Average Program Attendance
Description: Program attendance will be defined as average percentage of sessions attended by group.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Average percentage of sessions attended
Arm/Group | DPP-R | DPP-FB
Number analyzed (Participants) | 16 | 15
Average percentage of sessions attended | 69 (23.5) | 83 (26.6)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | DPP-R | DPP-FB
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT05387434/Prot_SAP_000.pdf